CLINICAL TRIAL: NCT04442659
Title: Prediction of Large Anterior Vessel Occlusion: a Prospective Observational Study Comparing Prehospital Prediction Scales
Brief Title: Prehospital Prediction of Large Anterior Vessel Occlusion
Acronym: PHPLAVO
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Alrijne Hospital (Other); Medical Center Haaglanden (Other); Haga Hospital (Other); Groene Hart Ziekenhuis (Other); Reinier de Graaf Groep (Other)
Responsible Party: Principal Investigator, NyikaKruyt, Md, PhD, Leiden University Medical Center
Other Study IDs: G18.058
Record Dates: First submitted 2020-06-15; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Stroke, Acute
Keywords: large vessel occlusion; Endovascular trombectomy; pre-hospital stroke triage
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pre hospital triage tool — EMS workers fill in an application containing 10-13 vclinical items

SUMMARY:
For the clinical benefit of intravenous thrombolysis "IVT" or intra-arterial thrombectomy "IAT" time is the most crucial factor. Reducing the time between stroke onset en treatment is therefore a major goal. Since IAT is only suitable for stroke due to large anterior vessel occlusion "LAVO" which is only performed in specialized comprehensive stroke centers "CSC", triage of LAVO-patients in the prehospital phase (i.e. in the ambulance) in order to directly allocate them to such a specialized CSC will save vital time (time=brain!). Several LAVO-prediction scales for clinical triage have been developed but most were tested in- hospital by experienced neurologists. Consequently, there is a great need for validation of these scales in the prehospital setting by Emergency Medical Services "EMS" personnel.

Objective: to recalibrate, validate performance and assess feasibility of several existing LAVO-prediction scales in the prehospital phase (i.e. assessment by EMS personnel).

Study design: multiregional, multicenter observational cohort study to investigate performance and feasibility of LAVO-prediction scales a.

Study population: all patients potentially eligible for IVTIAT according to the protocol used by EMS personnel except for when younger than 18 years.

DETAILED DESCRIPTION:
The study will be conducted in two EMS regions: Hollands Midden and Haaglanden. In addition, all hospitals in these regions that treat over 30 patients per year with IVT will participate, including at least 1 CSC with IAT-availability per region. These hospitals are: Leiden University Medical Center "LUMC"; Alrijne hospital (location Leiderdorp); Haaglanden Medical Center (HMC+); Haga hospital; LangeLand hospital (LLZ) and Reinier de Graaf hospital (RdGG).

The observational design is pragmatic and reflects standard practice for acute stroke care.

inclusion: All patients with suspected stroke potentially eligible for IVT/IAT as estimated by the on-site EMS nurse.

A web based application is used that merely structures observations that are currently noted on transport charts. EMS personnel will have access to the web-based application via the iPad/tablet/smartphone/computer on which the EMS transport chart is already filled out as part of standard care. Or via their patient record as used in the ambulance.

The application will consist of the following items:

* EMS transport number
* time of symptom onset
* probability of LAVO estimated by EMS nurse
* 9-12 questions to structure clinical observations made by the EMS nurse.

The application will be straightforward and designed in close co-operation with EMS personnel. With the items acquired all prediction scales can be reconstructed.

Data of the application will be retrieved retrospectively and coupled with retrospectively collected data from the participating hospitals by a trusted third party

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke code activated by EMS personnel

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All stroke codes within the ambulance regions of the Emergency medical services Hollands midden or Haaglanden.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
symptomatic Large Anterior Vessel Occlusion | on admission
  TICI score
Feasibility outcome | "within first hour"
  reconstruction rate of cuttoff and/or full scale

SECONDARY OUTCOMES:
final diagnosis | "Three months"
  diagnosis after discharge and/or after three months.
Endovascular therpay | "within first 24 hours of admission"
  EVT

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Stroke triage app — https://stroketriage.com/collect/start/16